CLINICAL TRIAL: NCT03744338
Title: Non-antibiotic Primary Prevention of Low Urinary Tract Infections: Evaluation of the Knowledge and Practices of Patients in the General Practitioner's Office, Observational and Descriptive Study in the Former Auvergne Region in France.
Brief Title: Prevention of Cystitis.
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-416
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Woman Aged 18 to 65
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — The questionnaire is composed of two parts:
  The first part let know the characteristics of the patients as age, the BMI, the socio-professional category, the current treatments, the medical-surgical antecedents of interest.

SUMMARY:
3436/5000 Urinary tract infections are a real public health issue. The frequency of these infections in France is estimated between 6 and 8 million in primary care (1) which represents 15% of antibiotics prescribed in primary care. Approximately 40-50% of women have had at least one UTI during their lifetime. (4) There is also an ecological issue by increasing the resistance of bacteria to antibiotics. (6) (7) The goal is to assess patients' knowledge and understandings to improve primary prevention.

The secondary objective will be to identify the demographic, sociological and ethiologic factors that may influence the knowledge and behavior of patients consulting in general medicine concerning means of prevention of cystitis.

This exploratory descriptive study is carried out on the basis of an anonymous questionnaire distributed in waiting rooms of GP offices after drawing lots in the former Auvergne region with prior approval of doctors. The inclusion criterion is to be a woman aged 18 to 65, consultant in general medicine.

24 general practitioners will be drawn in proportion to the distribution by department of the former region of Auvergne.

The primary outcome measure is to assess patients' knowledge and behaviors about how to prevent cystitis from responses to questionnaire items

. The duration of the study will be 6 weeks. The questionnaire consists of a section on the characteristics of patients including age, BMI, socio-professional category, current treatments, medico-surgical antecedents of interest and the other part consisting of 16 questions. on preventative measures to avoid cystitis with simple answers divided into "did you know" and "do it yourself", two questions about ecology and two other questions about lifestyle and other preventive practices.

It will also be collected data on the selected doctors: age, location, gynecological acts associated with general medicine.

The statistical analysis will be carried out with the software Stata . All statistical tests will be carried out at the risk of error of the first kind α of 5%. Patients will be described according to the variables: compliance with eligibility criteria, epidemiological characteristics, clinical characteristics and treatments. These analyzes will be complemented by the usual statistical tests, for example Chi2 test or Fisher-exact test for the comparison of categorical and anova variables or Kruskal-Wallis test if necessary for the quantitative variables. It seems difficult to propose for this exploratory observational study an estimate of the number of necessary subjects sufficiently robust and relevant. Nevertheless, it has been agreed to include at least 800 patients to establish possible specific profiles associated with patient knowledge and behavior The protocol, the information and consent form and the questionnaire were submitted for opinion to the Protection to Persons Committee.

DETAILED DESCRIPTION:
3436/5000 Urinary tract infections are a real public health issue. The frequency of these infections in France is estimated between 6 and 8 million in primary care (1) which represents 15% of antibiotics prescribed in primary care. Approximately 40-50% of women have had at least one UTI during their lifetime. (4) There is also an ecological issue by increasing the resistance of bacteria to antibiotics. (6) The goal is to assess patients' knowledge and understandings to improve primary prevention.

The secondary objective will be to identify the demographic, sociological and ethiologic factors that may influence the knowledge and behavior of patients consulting in general medicine concerning means of prevention of cystitis.

This exploratory descriptive study is carried out on the basis of an anonymous questionnaire distributed in waiting rooms of GP offices after drawing lots in the former Auvergne region with prior approval of doctors. The inclusion criterion is to be a woman aged 18 to 65, consultant in general medicine.

24 general practitioners will be drawn in proportion to the distribution by department of the former region of Auvergne.

The primary outcome measure is to assess patients' knowledge and behaviors about how to prevent cystitis from responses to questionnaire items

. The duration of the study will be 6 weeks. The questionnaire consists of a section on the characteristics of patients including age, BMI, socio-professional category, current treatments, medico-surgical antecedents of interest and the other part consisting of 16 questions. on preventative measures to avoid cystitis with simple answers divided into "did you know" and "do it yourself", two questions about ecology and two other questions about lifestyle and other preventive practices.

It will also be collected data on the selected doctors: age, location, gynecological acts associated with general medicine.

The statistical analysis will be carried out with the software Stata All statistical tests will be carried out at the risk of error of the first kind α of 5%. Patients will be described according to the variables: compliance with eligibility criteria, epidemiological characteristics, clinical characteristics and treatments. These analyzes will be complemented by the usual statistical tests, for example Chi2 test or Fisher-exact test for the comparison of categorical and anova variables or Kruskal-Wallis test if necessary for the quantitative variables. It seems difficult to propose for this exploratory observational study an estimate of the number of necessary subjects sufficiently robust and relevant. Nevertheless, it has been agreed to include at least 800 patients to establish possible specific profiles associated with patient knowledge and behavior The protocol, the information and consent form and the questionnaire were submitted for opinion to the Protection to Persons Committee.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 to 65, consultant in general medicine. (Any patient meeting the inclusion criteria may choose to answer the questionnaire in the waiting room of general practitioners selected by lot.)

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Woman aged 18 to 65
Sampling Method: Non-Probability Sample
Enrollment: 773 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Assessment of patients' knowledge and behaviors on means of prevention of cystitis from responses to questionnaire items | at 6 weeks
  The questionnaire is composed of two parts:
  The first part let know the characteristics of the patients as age, the BMI, the socio-professional category, the current treatments, the medical-surgical antecedents of interest.
  The other part consists of
  * 16 questions about preventative measures to avoid cystitis with simple answers divided into "did you know" and "do it yourself"
  * Two questions about ecology,
  * And two other questions about lifestyle and other preventive practices.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra CURINIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Francois M, Hanslik T, Dervaux B, Le Strat Y, Souty C, Vaux S, Maugat S, Rondet C, Sarazin M, Heym B, Coignard B, Rossignol L. The economic burden of urinary tract infections in women visiting general practices in France: a cross-sectional survey. BMC Health Serv Res. 2016 Aug 9;16(a):365. doi: 10.1186/s12913-016-1620-2. PMID 27507292
- [Background] Kunin CM. Urinary tract infections in females. Clin Infect Dis. 1994 Jan;18(1):1-10; quiz 11-2. doi: 10.1093/clinids/18.1.1. No abstract available. PMID 8054415
- [Background] Arpin C, Quentin C, Grobost F, Cambau E, Robert J, Dubois V, Coulange L, Andre C; Scientific Committee of ONERBA. Nationwide survey of extended-spectrum beta-lactamase-producing Enterobacteriaceae in the French community setting. J Antimicrob Chemother. 2009 Jun;63(6):1205-14. doi: 10.1093/jac/dkp108. Epub 2009 Mar 28. PMID 19329798